CLINICAL TRIAL: NCT02597257
Title: Efficacy and Safety of Lidocaine Infusion Treatment in Management of Neuropathic Pain: Randomized, Controlled, Comparative Study
Brief Title: Efficacy and Safety of Lidocaine Infusion Treatment in Management of Neuropathic Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Principal Investigator, Yong Chul Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1720150047
Record Dates: First submitted 2015-09-18; First posted 2015-11-05 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Postherpetic Neuralgia; Diabetic Polyneuropathy; Peripheral Neuropathy
Keywords: Lidocaine infusion therapy
MeSH Terms: conditions — Neuralgia, Postherpetic; Diabetic Neuropathies; Peripheral Nervous System Diseases | interventions — Lidocaine; Long-Term Synaptic Depression; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Saline (Placebo Comparator): * normal saline
  * total 250 ml
  * once a week
  * 4 times
  Interventions: Drug: Normal saline
- Lidocaine HCl (Active Comparator): * lidocaine 3 mg/kg mixed in normal saline
  * total 250 ml
  * once a week
  * 4 times
  Interventions: Drug: Lidocaine HCl

INTERVENTIONS:
Drug: Lidocaine HCl — lidocaine continuous infusion
  Other Names: 183903BIJ, Lidocaine HCl inj. 2% DAEHAN PHARM. CO., LTD.
  Arms: Lidocaine HCl
Drug: Normal saline — Normal saline continuous infusion
  Other Names: 228714BIJ, ISOTONIC SODIUM CHLORIDE DAEHAN PHARM. CO., LTD.
  Arms: Normal Saline

SUMMARY:
The investigators conducted a randomized, Double blind, and Controlled Study to evaluate the Efficacy and safety of Lidocaine Infusion Treatment in Management of Neuropathic pain.

DETAILED DESCRIPTION:
The investigators expect pain improvement after treatment with 3 mg/kg of lidocaine, continuously infused in normal saline 250 ml.

ELIGIBILITY:
Inclusion Criteria:

* postherpetic neuralgia, diabetic polyneuropathy, peripheral neuropathy
* NRS score > 4
* stable oral medication during the 1 month trial period
* volunteers with informed consent

Exclusion Criteria:

* pregnancy, breastfeeding, possibility of pregnancy
* pain from causes other than upper 3 indications
* hypersensitivity to lidocaine or other local anesthetics
* important disease of heart, kidney, liver or incurable disease that may affect the assessment of adverse effects, or may interfere with the completion of study
* severe conduction block
* history of other interventions that may affect the study
* Enrollment in other clinical trials within 30 days
* otherwise not suitable to study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
11-point Numeric Rating Scale | 1 week after the end of intervention
  Rating averaged daily pain score over a 7-day period, 0=on pain to 10=worst possible pain

SECONDARY OUTCOMES:
Brief Pain Inventory Short Form | at the end of intervention and 4 weeks after the end of intervention
  measurements of pain intensity, functionality, and impact of pain, rated on an 11-point Numerical Rating Scale (NRS) [0=no pain to 10=worst possible pain]
Shot Form McGill Pain Questionnaire | at the end of intervention and 4 weeks after the end of intervention
  15 pain descriptors ranked on a 4-stage intensity scale, the Present Pain Intensity index ranked on a 6-stage intensity and VAS (100-mm scale)
Patient Global Impression of Change | at the end of intervention and 4 weeks after the end of intervention
  7-point scale from very much improved to very much worse
Number of patients with grade 3 through grade 5 adverse events that are related to study drug, graded according to NCI CTCAE version 4.0 | through the study completion (7 weeks)
  AEs, laboratory values, vital signs, 12-lead ECG, finding from physical examination The intensity of AEs was graded according to the NCI common terminology criteria for adverse events v 4.0 on five point scale (grade 1 to 5: mild, moderate, severe, life-threatening and Death)
11-point Numeric Rating Scale | 4 weeks after the end of intervention
  Rating averaged daily pain score over a 7-day period, 0=on pain to 10=worst possible pain

CONTACTS AND LOCATIONS:
Overall Officials: Yong Chul Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Yong Chul Kim, Seoul, South Korea

REFERENCES:
- [Derived] Kim YC, Castaneda AM, Lee CS, Jin HS, Park KS, Moon JY. Efficacy and Safety of Lidocaine Infusion Treatment for Neuropathic Pain: A Randomized, Double-Blind, and Placebo-Controlled Study. Reg Anesth Pain Med. 2018 May;43(4):415-424. doi: 10.1097/AAP.0000000000000741. PMID 29381569